CLINICAL TRIAL: NCT03813667
Title: Palliative Care Coaching for Family Caregivers & Patients With Rare Advanced Lung Disease
Brief Title: Palliative Care Coaching for Families With Rare Advanced Lung Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Ubolrat Piamjariyakul, Associate Dean of Research, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1703528067
Record Dates: First submitted 2018-10-11; First posted 2019-01-23 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Lung Diseases; Rare Non-Neoplastic Disorder
Keywords: advanced lung diseases; Palliative Care; Dyspnea; pilot projects; Terminal Care
MeSH Terms: conditions — Lung Diseases; Dyspnea

STUDY DESIGN:
Intervention Model Description: This study uses a random control group comparison design to test the implementation of the FamPALcare intervention with R-ALD patients and their primary family caregivers.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care provider and outcome assessor including data collectors will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control patients have standard care given through the WVU hospital and outpatient clinics, prescribed by the patient's pulmonologist and recorded in the medical record
- Intervention (Experimental): The FamPALcare intervention group receives all standard care plus 2 weeks of home EOLPC coaching by community nurses experienced in end-of-life palliative care.
  Interventions: Behavioral: Intervention FamPALcare

INTERVENTIONS:
Behavioral: Intervention FamPALcare — The FamPALcare intervention includes all standard care information on R-ALD home care plus 2 weeks of EOLPC coaching by community nurses experienced in EOLPC. The nurse uses the "Conversation Ready" pamphlet to guide discussion of EOL preferences. The nurse will: (1) support the patient and family in making decisions about EOL care options based on their preferences; (2) discuss options for EOL care when the patient's R-ALD symptoms become severe; (3) encourage completion of the advance directive forms at next physician appointment. The nurse will use "teach-back" processes to ensure that FamPALcare discussions are clear.
  Other Names: FamPALcare
  Arms: Intervention

SUMMARY:
With one of the highest incidences of lung disease deaths in the nation, there is great need for home end-of-life palliative care in the rural, disadvantaged communities of West Virginia. The aims of this proposed study are to: (1) pilot test the nursing care intervention with patients and family members managing home supportive EOLPC for rare advanced lung disease and (2) collect research data to report in the NIH resubmission and future trials.

DETAILED DESCRIPTION:
Nearly 15 million Americans and greater than 10% of West Virginia (WV) residents live with and eventually die from Rare and Advanced Lung Diseases (R-ALD), including pneumoconiosis (i.e., dust, asbestos), and idiopathic pulmonary fibrosis. Patients with R-ALD experience refractory breathlessness, depression, fatigue, and extreme worry about their family members and cost of health care. With one of the highest incidences of lung disease deaths in the nation, there is great need for home EOLPC in the rural, disadvantaged communities of WV. The proposed EOLPC intervention (FamPALcare) is based on R-ALD experts' input, national EOLPC guidelines, and the PI's published EOLPC studies with breathlessness in end-stage heart failure (HF) patients.

This project is well-aligned with the National Institutes of Health (NIH) priority specific to "Appalachian populations experiencing extreme inequities and poor access to healthcare" and the NIH PAR on palliative care for family caregivers and patients with advanced lung diseases. The PI's NIH application review, which received a positive score, stated that this project will have a high impact on improving palliative care for rural families managing lung disease and the project can be translated to other rural communities. This is an initial study of coaching home-based palliative R-ALD care in rural Appalachia. The NIH review stated using the PI's culturally sensitive approaches for R-ALD was novel for chronic lung disease. Also, addressing both family caregivers' and patients' needs was noted as innovative and increased the potential for future funding, as was the rigorous protocol for observing intervention fidelity.

This study uses a random control group comparison design to test the implementation of the FamPALcare intervention with R-ALD patients and their primary family caregiver. Specific aims are to: (1) pilot test the FamPALcare nursing care intervention with patients and family members managing home supportive EOLPC for R-ALD and (2) collect research data to report in the PI's NIH resubmission and future trials. The control patients receive standard care given through the WVU hospital and outpatient clinics, prescribed by the patient's pulmonologist, and recorded in the medical record. The FamPALcare intervention group receives all standard care plus 2 weeks of home EOLPC coaching by community nurses experienced in EOLPC. Data will be collected at baseline, month one, and month three from patients and caregivers independently. This pilot study provides testing of our research guides and procedures that will be described to enhance the NIH resubmission and will determine power needed for the future RCT design.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with R-ALD, and their primary family caregivers dyad.
* All participants must be alert and oriented.
* Be able to read and write in English.

Exclusion Criteria:

* Patients who have received or are on a waiting list for a lung transplant
* Patients diagnosed with another terminal illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
patient outcomes | 3 months
  The intervention group R-ALD patients will report lower scores on breathlessness scale compared to control group patients at 3 months.
  Breathlessness is measured by Self-report shortness of breath scale (1 item, 0-10; 0-no shortness of breath, 10 = shortness of breath as bad as can be) (Gift, Narsavage, 1998

SECONDARY OUTCOMES:
family caregiver outcomes | 3 months
  The intervention group family caregivers will rate lower scores on Anxiety and Depression on PHQ-4 Scale compared to control group caregivers at 3 months.
  Anxiety and Depression are measured by PHQ-4 Scale, 4-item Likert scale.
patients' decision on EOLPC | 3 months
  The intervention group will report higher numbers of signed advance directives.
  This outcome is measured by the presence of signed advance directives in the medical record. Various types of advance directives will be identified.
Helpfulness of home R-ALD EOLPC intervention | 3 months
  Each patient and family member will rate the 11-item Likert Intervention on the Helpfulness scale at 3 months. Range 1-5, 1= strongly disagree/not helpful and 5 = strong agree/helpful.

CONTACTS AND LOCATIONS:
Overall Officials: Ubolrat Piamjariyakul, PhD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University Hospital, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot RCT, the researchers do not want to share the IPD.

REFERENCES:
- [Derived] Piamjariyakul U, Smothers A, Young S, Petitte T, Wen S, Morrissey E, Shafique S, Zulfikar R, Sangani R, Smith CE. Palliative care for rare advanced lung diseases in underserved Appalachia: Study protocol for a randomized controlled trial. J Adv Nurs. 2020 Aug;76(8):2182-2190. doi: 10.1111/jan.14395. Epub 2020 May 2. PMID 32297352